CLINICAL TRIAL: NCT04903873
Title: An Open-Label, Phase 1/2 Study to Evaluate Safety, Efficacy, and Pharmacokinetics of EU101, an Agonistic Anti-CD137 (4-1BB) Monoclonal Antibody in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate Safety, Efficacy, and Pharmacokinetics in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eutilex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EU-CTS101-I-01
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor; Renal Cell Cancer Metastatic; Non-Small Cell Lung Cancer; Renal Cell Carcinoma; Prostate Cancer
Keywords: Renal Cell Carcinoma; Prostate Cancer; Dose Escalation; Maximum tolerated dose
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EU101: Dose Escalation Cohort (Experimental): Participants with advanced solid tumors will receive EU101 intravenously once every 3 weeks (3 weeks = 1 cycle) with escalating doses starting from 0.05 milligrams per kilogram (mg/kg) to 10 mg/kg until disease progression, unacceptable toxicities or death, withdrawal of consent, end of study, or physician's decision, whichever occurs first.
  Interventions: Drug: EU101
- EU101: Dose Expansion Cohort 1 (Experimental): Participants with CRC will receive EU101 intravenously once every 3 weeks (3 weeks = 1 cycle) with a determined recommended phase 2 dose until disease progression, unacceptable toxicities or death, withdrawal of consent, end of study, or physician's decision, whichever occurs first.
  Interventions: Drug: EU101
- EU101: Dose Expansion Cohort 2 (Experimental): Participants with NSCLC will receive EU101 intravenously once every 3 weeks (3 weeks = 1 cycle) with a determined recommended phase 2 dose until disease progression, unacceptable toxicities or death, withdrawal of consent, end of study, or physician's decision, whichever occurs first.
  Interventions: Drug: EU101

INTERVENTIONS:
Drug: EU101 — EU101 will be administered via intravenous infusion.

SUMMARY:
Phase 1 (Dose Escalation) of this study will assess the safety, tolerability, dose-limiting toxicity (DLT), and will determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of EU101 in participants with advanced solid tumors. Phase 2 (Dose Expansion) of the study will assess the antitumor effect of EU101 in two indications including colorectal cancer (CRC) and non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic or locally advanced solid tumors for which no standard therapy exists or standard therapy has failed because of disease progression or unacceptable toxicities. Also includes patients who cannot be treated with standard therapy because of underlying/existing medical condition.
* Cohort 1 (colorectal cancer): a) CRC (including microsatellite instability-high [MSI-H] and microsatellite-stable [MSS]) regardless of RAS mutation. b) Disease progression within 3 months after last administration of approved standard therapies. c) Prior cytotoxic chemotherapy for metastatic disease include all the following agents: fluoropyrimidine, oxaliplatin, and irinotecan
* Adjuvant chemotherapy-based treatments count as prior therapy, as long as relapse had occurred within 6 months of completion of such therapies, prior anti-epidermal growth factor receptor (EGFR) therapy (cetuximab, panitumumab), anti-angiogenic therapy (bevacizumab, aflibercept, ramucirumab), regorafenib, and TAS-102 are allowed. d) No more than 5 prior therapies for metastatic disease. For participants who had disease recurrence within 6 months of completing adjuvant chemotherapy, the adjuvant regimen can be considered as 1 chemotherapy regimen for metastatic disease
* Cohort 2 (NSCLC): a) NSCLC without known EGFR, anaplastic lymphoma kinase (ALK), and ROS1 genomic tumor aberrations. b) No standard therapy exists or standard therapy has failed. c) No more than 3 prior therapies for metastatic disease
* Phase 2: At least 1 measurable lesion per RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2
* Adequate organ and bone marrow function (Hemoglobin >9.0 g/dL, Absolute neutrophil count ≥1,500/μL, Absolute lymphocyte count ≥600 and ≤2,500/μL, Platelet count ≥100,000/μL, Total bilirubin ≤1.5 × upper limit of normal, Alanine aminotransferase and aspartate aminotransferase ≤2.5 × ULN, Serum creatinine ≤1.5 × ULN or creatinine clearance >30 mL/min, Prothrombin time and activated partial thromboplastin time ≤1.5 × ULN)
* Life expectancy of at least 12 weeks
* Voluntarily provided a written consent to participate in the study
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within the 7 days before study drug administration
* WOCBP and sexually active fertile male patients with partners who are WOCBP must agree to use 2 highly effective methods of contraception throughout the course of the study and for 12 weeks after the last dose of study drug.

Key Exclusion Criteria:

* Primary central nervous system (CNS) tumor (Phase 1), CNS metastasis, and/or carcinomatous meningitis. Participants with prior brain metastases treated at least 4 weeks before the first dose of EU101 that are clinically stable and do not require chronic corticosteroid treatment are allowed. Untreated but asymptomatic and clinically stable brain metastases per investigator's discretion are allowed
* Received prior therapy with any anti-CD137 monoclonal antibody (mAb) or agent
* Major surgery requiring general anesthesia within 3 weeks before first dose of EU101 or still recovering from prior surgery
* Active infection that is not controlled or requires intravenous antibiotics in the last 2 weeks
* History of allogeneic tissue or organ transplant
* Active hepatitis B virus or hepatitis C virus infection
* History of any noninfectious hepatitis
* Human immunodeficiency virus (HIV) infection
* Received or receiving systemic corticosteroid therapy or any other form of systemic immunosuppressive medicaion 1 week before first dose of EU101
* Known severe (≥Grade 3) hypersensitivity reactions to antibody, or severe reaction to immuno-oncology agents requiring treatment with steroids
* Konwn or suspected hypersensitivity to EU101 or any component of its formulation
* Current or history of interstitial lung disease, anaphylaxis, uncontrolled asthma, or pneumonitis that has required systemic corticosteroids
* Patients with second primary cancer
* Clinically significant concurrent cardiovascular disease
* Pregnant women, breasfeeding women, WOCBP, or men with partners who are WOCBP who do not agree to use adequate contraceptive measures
* Determined as unable to participate in the study per investigator's judgment

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants With Adverse Event (AEs) and Serious Adverse Events (SAEs) and Adverse Events Leading to Discontinuation | Baseline up to 30 months
Phase 1: Number of Participants With Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (Each cycle is of 21 Days)
Phase 1: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters | Baseline up to 24 months
  Laboratory assessments include hematology, serum chemistry, other blood tests, coagulation, and urine analysis. Number of participants with clinically significant abnormalities will be reported.
Phase 1: Number of Participants With Clinically Significant Abnormalities in Vital Signs | Baseline up to 24 months
  Vital signs will include body temperature, pulse rate, and systolic and diastolic blood pressure measurements. Number of participants with clinically significant abnormalities will be reported.
Phase 1: Number of Participants With Clinically Significant Abnormalities in Physical Examination | Baseline up to 24 months
  Physical examination will include head, eyes, ears, nose and throat; heart; lungs; abdomen; skin; cervical and axillary lymph nodes; and neurological and musculoskeletal systems. Number of participants with clinically significant abnormalities will be reported.
Phase 1: Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) | Baseline up to 24 months
  ECG parameters included heart rhythm, pulse rate intervals, QRS, QT intervals, RR intervals and corrected QT(QTc) intervals. Number of participants with clinically significant abnormalities will be reported.
Phase 2: Objective Response Rate (ORR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Objective response rate (ORR), defined as the percentage of participants with a best overall response (BOR) of either a complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for solid tumors by investigators.

SECONDARY OUTCOMES:
Phase 1: Objective Response Rate (ORR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Objective response rate (ORR), defined as the percentage of participants with a BOR of either a complete response (CR) or partial response (PR), per RECIST version 1.1 for solid tumors by investigators.
Phase 1 and 2: Duration of Response (DOR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 56 months)
Phase 1 and 2: Disease Control Rate (DCR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 56 months)
  DCR will be defined similarly to ORR but also including stable disease (SD) in the categorization of response (i.e, RECIST response of either CR, PR, or SD).
Phase 1 and 2: Time to Response (TTR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 56 months)
Phase 1 and 2: Time to Progression (TTP) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 56 months)
Phase 1 and 2: Durable Clinical Benefit (DCB) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 56 months)
  DCB will be defined similarly to DCR but additionally specifying that the disease control be achieved for at least 12 weeks consecutive (i.e, RECIST response of CR, PR or SD for greater than or equal to [>=] 12 weeks consecutive).
Phase 1 and 2: Progression-Free Survival (PFS) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 56 months)
Phase 1 and 2: Overall survival (OS) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 56 months)
Phase 1 and 2: Maximum Observed Serum Concentration (Cmax) of EU101 | Cycle 1: Pre-dose up to 336 hours post-dose; Cycle 2: 504 hours post-dose; Cycle 3: Pre-dose (Each cycle is of 21 days)]
  Cmax is defined as maximum observed serum concentration.
Phase 1 and 2: Trough Serum Concentration (Ctrough) of EU101 | Cycle 1: Pre-dose up to 336 hours post-dose; Cycle 2: 504 hours post-dose; Cycle 3: Pre-dose (Each cycle is of 21 days)]
  Ctrough is steady-state pre-dose concentration.
Phase 1 and 2: Time to Reach Maximum Observed Serum Concentration (Tmax) of EU101 | Cycle 1: Pre-dose up to 336 hours post-dose; Cycle 2: 504 hours post-dose; Cycle 3: Pre-dose (Each cycle is of 21 days)]
  Tmax is defined as time to reach maximum observed serum concentration.
Phase 1 and 2: Area Under the Serum Concentration-Time Curve From Time Zero to 24 Hours Post-dose (AUC0-24) of EU101 | Cycle 1: Pre-dose up to 336 hours post-dose; Cycle 2: 504 hours post-dose; Cycle 3: Pre-dose (Each cycle is of 21 days)]
  AUC0-24 is defined as the area under the serum concentration versus time curve from time zero (pre-dose) to 24 hours post-dose (0 to 24).
Phase 1 and 2: Area Under the Serum Concentration-Time Curve From Time Zero to the Last Measurable Concentration (AUC0-last) of EU101 | Cycle 1: Pre-dose up to 336 hours post-dose; Cycle 2: 504 hours post-dose; Cycle 3: Pre-dose (Each cycle is of 21 days)]
  AUC0-last is defined as area under the serum concentration time-curve from time zero to the time of last measured concentration.
Phase 1 and 2: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of EU101 | Cycle 1: Pre-dose up to 336 hours post-dose; Cycle 2: 504 hours post-dose; Cycle 3: Pre-dose (Each cycle is of 21 days)]
  AUCinf is defined as area under the serum concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Phase 1 and 2: Elimination Half-Life Time (T1/2) of EU101 | Cycle 1: Pre-dose up to 336 hours post-dose; Cycle 2: 504 hours post-dose; Cycle 3: Pre-dose (Each cycle is of 21 days)]
  T1/2 is defined as plasma decay half-life is the time measured for the serum concentration to decrease by one half.
Phase 1 and 2: Apparent Volume of Distribution (Vd/F) of EU101 | Baseline (Day 1)
  Vd/F is defined as volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug.
Phase 1 and 2: Apparent Oral Clearance of (CL/F) of EU101 | Baseline (Day 1)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Phase 1 and 2: Mean Residence Time (MRT) of EU101 | Baseline (Day 1)
  MRT is defined as AUMC(0 - inf) divided by AUC(0 - inf), where AUMC(0 - inf) is the area under the first moment curve from time 0 extrapolated to infinite time.
Phase 1 and 2: Renal clearance (CLr) of EU101 | Baseline (Day 1)
  CLr is defined as renal clearance is the volume of plasma completely cleared of EU101 by the kidneys per unit time.
Phase 1 and 2: Number of Participants with Positive Antidrug Antibodies (ADA) | Baseline up to 56 months
  The immunogenic potential of EU101 will be assessed by summarizing the number of participants who develop detectable antidrug antibody (ADAs).
Phase 2: Number of Participants With AEs and SAEs by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Time from first dose of study treatment up to 30 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley Center, Dallas, Texas
- South Korea (4):
  - National Cancer Center, Ilsan
  - Samsung Seoul Hospital, Seoul
  - Seoul Asan, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No